CLINICAL TRIAL: NCT04682743
Title: Efficacy of Ondansetron Versus Paracetamol for Prevention of Post-Operative Shivering
Brief Title: Prevention of Post-Operative Shivering
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-122-2020
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Post-Operative Shivering
MeSH Terms: interventions — Acetaminophen; Ondansetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- saline group (Sham Comparator)
  Interventions: Drug: normal saline
- ondansetron group (Active Comparator)
  Interventions: Drug: ondansetron
- paracetamol group (Active Comparator)
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: paracetamol — received intravenous one gram of paracetamol over a 15-minute period,
  Arms: paracetamol group
Drug: ondansetron — received intravenous 8 mg of ondansetron over a 15-minute period.
  Arms: ondansetron group
Drug: normal saline — received intravenous 0.9% normal saline over a 15-minute period.
  Arms: saline group

SUMMARY:
Shivering and vasoconstriction are thermoregulatory mechanisms that are required to increase core body temperature (BT) in patients with core hypothermia.

paracetamol is an antipyretic drug that has been in clinical use for a long time.

It can lower the BT of febrile and nonfebrile patients. A previous study demonstrated that orally administered paracetamol can suppress in a dose-dependent manner the increase in the BT of patients with acute ischemic stroke. However, few studies have evaluated the effects of paracetamol on postoperative shivering.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18-40 years.
* ASA physical status I and II
* Both genders
* Patients scheduled for elective mega-liposuction surgery under combined general epidural anesthesia

Exclusion criteria

* Patients who refused to participate in the study,
* ASA physical status more than II,
* any contraindications to regional anesthesia,
* surgical duration less than two hours or exceeding six hours,
* giving history of any of the following; allergy to the study medications used, system impairment, alcohol abuse, any endocrine disease affecting body temperature such as thyroid disorders,
* any psychiatric or neurological disorders, convulsions, patient receiving vasodilators or medications likely to alter thermoregulation,
* Finally if their body temperature was recorded to surpass 37.5ºC or <36.5°C before enrolment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Incidence of shivering | UP TO 1 HOURE
  60 min postoperatively

SECONDARY OUTCOMES:
The assessment the core temperatures | UP TO 24 HOURE
  temperatures
postoperative shivering scores | up to 2 hours
  "0" indicated no shivering; "1," piloerection or peripheral vasoconstriction, but no visible shivering; "2," muscular activity in only 1 muscle group; "3," muscular activity in >1 muscle group, but not generalized; and "4," shivering involving the whole body.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided